Global Clinical Development Template CCD-6230.T01 Revision 01



# Statistical Analysis Plan

| Protocol Number/version | DBC-18PENDL01/Version 3.0 06Feb2019 |
|---|---|
| Protocol Title | Comparative User Experiences with BD Nano™PRO 32G Extra Thin Wall |
| | Pen Needle vs the Terumo Nanopass® 34G Pen Needle |
| SAP Date | February 20, 2019 |
| Version History | Version 2.0 20Feb2019 Administrative change (Protocol version updated) |
| | Version 1.0 24Jan2019 Original Release |

THIS DOCUMENT IS PROPRIETARY TO BECTON DICKINSON. NO PART OF IT MAY BE DISTRIBUTED OR SHARED WITH PERSONS OTHER THAN BD ASSOCIATES WITHOUT WRITTEN PERMISSION FROM GLOBAL CLINICAL DEVELOPMENT (GCD).

# Approval

| Function | Name | Signature |
|---|---|---|
| Study Statistician (Author) | Wen Yue | This document is signed electronically in the eTMF system. |
| Medical Affairs Team<br>Representative | Shahista Whooley | This document is signed electronically in the eTMF system. |
| Study Manager | Jonathan<br>Washington | This document is signed electronically in the eTMF system. |
| Associate Director, Statistics | Julie Bérubé | This document is signed electronically in the eTMF system. |

DBC-18PENDL01 




# Contents

| 1 | List of Abbreviations and Definitions |
|---|---|
| 2 | Overall Study Description 2.1 Study Background 2.2 Study Objectives 2.3 Study Design 2.4 Endpoints 2.4.1 Primary Endpoints 2.4.2 Secondary Endpoints 2.4.3 Exploratory Endpoints 2.4.4 Safety Endpoints 2.5 Acceptance Criteria 2.5.1 Primary Objective 2.5.2 Secondary Objectives 2.5.3 Exploratory Objectives |
| 3 | Sample Size |
| 4 | Intended Statistical Software |
| 5 | Data 5.1 Database Information |
| 6 | Statistical Analysis / Calculations 5.1 Derived Variables |
| 7 | Safety Analysis |
| 8 | Example Reports 8.1 Study Execution 8.1.1 Analysis Population Set(s) 8.1.2 Data Exclusions 8.1.3 Executive Summary |

DBC-18PENDL01



| | 8.2 | Analysis and Results | 6 |
|---|-----|-----------------------------------|---|
| | | 8.2.1 Injection Pain | 6 |
| | | 8.2.2 Injection force | 8 |
| | | 8.2.3 Needle Bending | 9 |
| | | 8.2.4 Leakage from Injection Site | 9 |
| | | 8.2.5 Exploratory Objectives | 1 |
| | 8.3 | Demographics and Diabetes History | 1 |
| 9 | App | pendix 2 | 3 |
| | 9.1 | Discontinued Data | 3 |
| | 9.2 | Missing Data | 3 |
| | 9.3 | Adverse Events | 3 |

DBC-18PENDL01 



# 1 List of Abbreviations and Definitions

- **AE:** Adverse event
- **BD:** Becton Dickinson and Company
- GCD: Global Clinical Development, BD
- CI: Confidence Interval
- CRF: Case Report/Record Form
- **G**: Gauge
- **IFU:** Instruction for Use
- NI: Non Inferiority
- VAS: Visual Analog Scale
- RS: Randomization schedule
- SAE: Serious Adverse Event
- SAP: Statistical Analysis Plan
- **SD:** Standard Deviation

DBC-18PENDL01 



# 2 Overall Study Description

# 2.1 Study Background

Pen needles are a component of pen-based injection systems routinely utilized for parenteral administration of medicaments such as insulin. In 2010, BD introduced a 4mm x 32G pen needle. At that time it was the shortest and thinnest pen needle available. In addition to lowering the risk for intramuscular injections, this pen needle was demonstrated to be preferred by patients vs. their current pen needles. Since its introduction, competitors have launched similar length pen needles with thinner gauge needles, such as 33G and 34G. The intent of this comparative use study is to determine whether patient experiences are different when using the BD Nano™ PRO 4mm x 32G extra thin wall, 5-bevel pen needle (herein referred to as BD Nano™ PRO) vs the Terumo Nanopass® 4mm x 34G (thinner gauge) pen needle (herein referred to as Terumo Nanopass®). These experiences include injection pain, force to deliver dose, bending, and ability to deliver full dose (leakage).

# 2.2 Study Objectives

#### • Primary Objective

Demonstrate non-inferiority of the BD Nano<sup>™</sup> PRO pen needle compared to the Terumo Nanopass<sup>®</sup> pen needle for injection pain.

#### • Secondary Objectives

Demonstrate superiority of BD Nano<sup>™</sup> PRO vs Terumo Nanopass<sup>®</sup> pen needle for the following:

- 1. Leakage from the needle tip and the injection site (measurements combined) after removal from body
- 2. Subject perceived force required to deliver dose
- 3. Patient end needle bending after removal from body
- 4. If primary outcome demonstrates non-inferiority then evaluate for superiority of Nano™PRO vs Terumo Nanopass®

#### • Exploratory Objectives

Compare BD Nano<sup>™</sup> PRO vs Terumo Nanopass<sup>®</sup> for the following:

- 1. Injection time
- 2. Patient end needle breaking at any time
- 3. Survey responses pertaining to subjective assessments of pen needle characteristics

DBC-18PENDL01 



# 2.3 Study Design

This is a subject partially blinded, block randomized, prospective, single-visit, multi-center study to compare user experiences with BD Nano™ PRO pen needle vs. the thinner commercially available Terumo Nanopass® pen needle. The study will include a minimum of 55 Japanese American study subjects having Type 1 or Type 2 diabetes. Study conduct will consist of one 60 to 120 minute Site visit in which pre-set doses of saline will be abdominally delivered by subjects via a reusable insulin pen device. All pen needles will be attached by Study Staff and pen needle outer cover and inner shield will be removed for subjects. Subjects are to perform 12 injections into the abdomen (6 pairs of injections). Pairs of injections will be evaluated and each pair will contain one BD Nano™ PRO and one Terumo Nanopass® pen needle. Subjects will not see pen needle labels or be informed which pen needle is being used to inject. The BD Nano™ PRO has a distinct configuration and subjects will most likely notice the difference vs the Terumo Nanopass®. Subjects will not be informed of the Terumo Nanopass® brand, length or gauge. The pen needle order within the pairs of injections will be randomized for each subject and the pairs will be randomized to various abdominal injection sites within each subject. Besides being informed of the requirement to insert the pen needles 'straight-in' (perpendicular), subjects will be instructed to use their usual injection technique.

## 2.4 Endpoints

#### 2.4.1 Primary Endpoints

**Injection Pain**: Each Subject will evaluate pain after completion of each pair of injections using a 15 cm relative Visual Analog Scale (VAS).

#### 2.4.2 Secondary Endpoints

After each injection:

- Leakage: After saline delivery equivalent to 30U of U100 insulin (0.3mL) and Subject removal of pen needle from body, Study Staff will use the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage.

  Leakage will be considered to be present if measurement is equivalent to or greater than 5% of dose (equivalent to or greater than 1.5U of U100 insulin equivalent to ≥ 0.015g).
- Needle bending: Study Staff will use a provided needle bend scale and visually inspect retained pen needles to determine the presence of bending. If present, study staff will determine and document degree of bend with the provided scale. For the purpose of answering the study objective, needle bend will be considered equivalent to or greater than 2 on the bend rating scale.

After each pair of injections:

• Injection force: Each Subject will evaluate perceived injection force after each pair of injections using a 5-point Likert scale (from 1st injection required much less force to deliver medication to 2nd injection required much less force to deliver medication).

DBC-18PENDL01 



#### 2.4.3 Exploratory Endpoints

During each injection: Injection time - includes the following time periods for each injection

- Time from when subject first pushes injection button to time button fully depressed (delivery time)
- Time from when injection button fully depressed to when pen needle removed from body
- Total injection time the 2 time periods above combined (total injection time)

#### After each injection:

• Breaking: Study Staff will record any patient end needle breakage. Breakage is defined as the patient-end metal cannula separated into two pieces.

#### After all injections completed:

- Survey responses: Subject completes a 5-point Likert scale survey (from Disagree to Agree). Subject will be instructed to respond to the questions based on their usual (in-home use) injection experience. Subject responses to survey questions will be tallied. The survey includes the following four questions:
  - 1. Injection pain affects my level of satisfaction with my treatment.
  - 2. Injection pressure needed to deliver the dose affects my level of satisfaction with my treatment.
  - 3. Post injection leakage increases my level of concern that I may not be receiving my full dose of medication.
  - 4. A bent needle increases my level of concern about the reliability of my injection.

## 2.4.4 Safety Endpoints

Occurrence of adverse events will be evaluated, recorded, and followed up as required.

#### 2.5 Acceptance Criteria

#### 2.5.1 Primary Objective

BD Nano<sup> $\mathbb{M}$ </sup> PRO non-inferior to Terumo Nanopass<sup> $\mathbb{R}$ </sup> for injection pain with partially blinded injections based on relative VAS, where -75mm indicates worse pain for BD Nano<sup> $\mathbb{M}$ </sup> PRO and +75mm indicates worse pain for Terumo Nanopass<sup> $\mathbb{R}$ </sup> with a non-inferiority criterion of -10mm.

#### 2.5.2 Secondary Objectives

- The BD Nano<sup>™</sup> PRO will be evaluated for superiority vs Terumo Nanopass<sup>®</sup> for leakage, injection force, and bending.
- If the BD Nano<sup>™</sup> PRO demonstrates non-inferiority for injection pain for the Primary Objective, compare the BD Nano<sup>™</sup> PRO vs Terumo Nanopass<sup>®</sup> for superiority.

DBC-18PENDL01 



#### 2.5.3 Exploratory Objectives

No formal acceptance criterion has been established for the following objectives - time to deliver dose, total injection time, and survey responses after all injections completed.

# 3 Sample Size

Leakage data is currently being used to calculate sample size.

Based on previous study data (BDT-2P00116) where leakage is equal to or greater than 1.5U was observed in 20/298 (6.7%) of injections performed with Terumo Nanopass<sup>®</sup> and in 3/297 (1%) of injections performed with BD Nano<sup>™</sup> PRO, a simulation was performed (code found in SVN repository under DBC-18PENDL01Size Bayesian prior proportion.R) indicating that 292 injections per each pen needle type would provide 90% power to show BD Nano<sup>™</sup> PRO superiority to Terumo Nanopass<sup>®</sup>. If each Subject tests 6 pairs of pen needles, 292 injections per each pen needle requires 49 subjects (rounded to 50 subjects). 50 Subjects will generate data for 600 pen needles: 300 pen needle pairs - 300 BD Nano<sup>™</sup> PRO and 300 Terumo Nanopass<sup>®</sup>. A 10% buffer was added (to compensate for subject attrition or unusable data), leading to a planned enrollment number of 55 subjects.

Pain: Assuming the SD for relative VAS is around 50mm (based on DBC-17NUCLS07), a sample size of 300 pairs (50 Subjects x 6 pairs) has >90% power of passing a -10mm NI criteria, assuming a true average of -0.5mm in favor of Terumo Nanopass® (based on a 2-sided 95% CI for the mean).

#### 4 Intended Statistical Software

This document was generated with R version 3.5.1 (2018-07-02) and the following packages (version) were used: assertthat (0.2.0), base (3.5.1), BDbasics (0.2.4), bindr (0.1.1), bindrcpp (0.2.2), colorspace (1.3.2), compiler (3.5.1), crayon (1.3.4), datasets (3.5.1), dplyr (0.7.6), ggplot2 (3.0.0), glue (1.3.0), graphics (3.5.1), grDevices (3.5.1), grid (3.5.1), gtable (0.2.0), lattice (0.20.35), lazyeval (0.2.1), magrittr (1.5), methods (3.5.1), munsell (0.5.0), nlme (3.1.137), pillar (1.3.0), pkgconfig (2.0.2), plyr (1.8.4), purrr (0.2.5), R6 (2.2.2), Rcpp (0.12.18), reshape2 (1.4.3), rJava (0.9.10), rlang (0.2.2), scales (1.0.0), stats (3.5.1), stringi (1.1.7), stringr (1.3.1), tibble (1.4.2), tidyselect (0.2.4), tools (3.5.1), utils (3.5.1), withr (2.1.2), xlsx (0.6.1), xlsxjars (0.6.1), xtable (1.8.3).

The study will be conducted within the same environment or more recent versions.

## 5 Data

#### 5.1 Database Information

The input data will consist in several csv (comma separated values) files exported from Clindex.

Files will be saved in

https://svn.bdx.com:8443/svn/stats\_and\_dm/DM and Stats Outputs/DBC/DBC-18PENDL01/Data and read directly into R for analysis.

DBC-18PENDL01 



# 5.2 Analysis Population Set(s)

All data collected will be analyzed and reviewed for possible exclusion based on significant outliers or protocol deviations.

Injections where bleeding was observed will not be used in the leakage analyses.

Analyses of relative data will only include pairs where both injections were completed.

Demographic information and Diabetes history collected for all subjects randomized will be tabulated.

Data from all subjects will be included in the summary of safety parameters.

# 6 Statistical Analysis / Calculations

#### 6.1 Derived Variables

# 6.1.1 Relative VAS Scale

After completion of each pair of injection, subjects will be asked to compare pain between the pen needles using a 150mm relative VAS Scale. Marks made on the 150mm relative VAS Scale are read using a 0 - 20 grid and the resulting discrete scores entered into the database. The results will be transformed to a [-75mm, 75mm] scale for analysis and reporting, where positive scores will reflect less pain for BD Nano Pro and negative scores will reflect less pain for Terumo.

Subjects will draw a vertical line on a relative VAS scale for each pair of injections, to indicate their relative pain perception for the pen needle used first or second in the pair. A vertical line drawn to the left of the center mark indicates that the 1st injection was less painful. A vertical line drawn to the right of the center mark indicates that the 2nd injection was less painful. A vertical line drawn at the center mark indicates no difference. Figure 1 shows an example of a 150mm (may not be to scale) relative VAS scale.

The scores are entered into the database on a discrete 0-20 scale. These scores will be transformed to a 150mm VAS on a [-75mm, 75mm] scale as follows:

Let  $Y_{recorded}$  (= 0, 1,  $\cdots$ , 20) be the recorded VAS score, the first transformation for the analysis of VAS score,  $Y_{analysis}^*$  (mm), will be calculated as:

$$Y_{analysis}^* = \frac{150}{20} * Y_{recorded} - 75 \tag{1}$$

The sign of the VAS responses  $Y_{analysis}^*$  will then be adjusted depending on which pen needle was used in the first and in the second injection, so that positive scores (+) will reflect less pain for BD Nano and negative scores (-) will reflect less pain for Terumo. Let  $Y_{analysis}$  be the final relative VAS score used for the analysis. Then:

$$Y_{analysis} = \begin{cases} Y_{analysis}^*, & \text{if BD Nano is provided in the 2}^{\text{nd}} & \text{injection} \\ -Y_{analysis}^*, & \text{if BD Nano is provided in the 1}^{\text{st}} & \text{injection} \end{cases}$$
(2)

DBC-18PENDL01 



Which injection was less painful?



Figure 1: VAS Scale for Injection Pain

#### 6.1.2 Leakage Scale

Study Staff will use the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage. Leakage will be considered to be present if measurement is equivalent to or greater than 5% of dose (equivalent to equal to or greater than 1.5U of U100 insulin (or 0.015g)). A binary leakage variable will be created with the equation below:

$$Y_{Leakage} = \begin{cases} \text{Yes, if recorded leakage} \ge 0.015g\\ \text{No, if recorded leakage} < 0.015g \end{cases}$$
(3)

DBC-18PENDL01 



# 6.1.3 Injection force

Injection force will be evaluated after each pair of injections using a 5-point Likert scale and the results will be converted to ratings of -2 to 2 as below:

$$Y_{Injectionforce}^* = \begin{cases} -2, & \text{if 1st injection significantly less thumb force} \\ -1, & \text{if 1st injection slightly less thumb force} \\ 0, & \text{if no difference} \\ 1, & \text{if 2nd injection slightly less thumb force} \end{cases} \tag{4}$$

The sign of the injection force responses  $Y_{Injectionforce}^*$  will then be adjusted depending on which pen needle was used in the first and in the second injection, so that positive scores (+) will reflect less thumb force for BD Nano and negative scores (-) will reflect less thumb force for Terumo. Let  $Y_{Injectionforce}$  be the final injection force score used for the analysis. Then:

$$Y_{Injectionforce} = \begin{cases} Y_{Injectionforce}^{*}, & \text{if BD Nano is provided in the 2}^{\text{nd}} & \text{injection} \\ -Y_{Injectionforce}^{*}, & \text{if BD Nano is provided in the 1}^{\text{st}} & \text{injection} \end{cases}$$
(5)

The responses will also be converted to 3 categories: favoring Terumo Nanopass<sup>®</sup> (negative ratings), no difference (0 ratings) and favoring BD Nano<sup>TM</sup> PRO (positive ratings) with the equation below:

$$Y_{Injectionforce(categorical)} = \begin{cases} \text{Terumo with less injection force if recorded rating } < 0 \\ \text{No difference, if recorded rating } = 0 \\ \text{BD Nano with less injection force if recorded rating } > 0 \end{cases}$$
 (6)

DBC-18PENDL01 



# 6.2 Analysis Method

This section provides a detailed description of the statistical analysis that will be performed in this study.

Unless otherwise stated, all the statistical tests are two-sided at a significance level of 5%.

Summary statistics (number of observations, mean, 95% CI for mean, median, standard deviation and range) for all quantitative responses will be presented in tables. Frequency tables with number of observations, percentage of total will be created for all discrete responses.

Bar plots may be provided for some responses.

#### 6.2.1 Analysis of Injection pain

A two-sided 95% confidence intervals will be calculated for the average rating. A modeling approach will be used to adjust for the pair order effect, BD order effect within pair (due to the often-observed bias towards favoring the last pen needle used in a pair), abdomen site effect and random subject effect. Results will be tested for non-inferiority, followed by superiority:

- If the lower bound of the CI is > -10mm, we can conclude in non-inferiority.
- If the lower bound of the CI is > 0mm, we can conclude in superiority.

DBC-18PENDL01 



```
> ## Example for estimated pen needle subgroup means
> ## if the lower CL is > -10, non-inferiority is satisfied
> ## if the lower CL is > 0, superiority is satisfied
> library(emmeans)
> emmeans(model.fit, ~1)
```

```
1 emmean SE df lower.CL upper.CL overall 24.10616 3.666296 145.14 16.85993 31.35238
```

Degrees-of-freedom method: kenward-roger

Confidence level used: 0.95

#### 6.2.2 Analysis of Injection force

The responses in 5-point Likert scale will be converted to ratings of -2 to 2 (where positive ratings favor BD, see section 6.1.3) and a two-sided 95% confidence interval will be calculated for the average rating. If the lower bound of the CI is > 0, we can conclude in superiority. A modeling approach will be used to adjust for the pair order effect, BD order effect within pair, abdomen site effect and random subject effect.

Responses will also be converted to 3 categories: favoring Terumo Nanopass<sup>®</sup> (negative ratings), no difference (0 ratings) and favoring BD Nano<sup>™</sup>PRO (positive ratings) (see Section 6.1.3). The difference in percentage of responses with a preference for BD Nano vs Terumo Nanopass will be calculated by Bayesian approach, adjusting for the "no preference" category.

#### 6.2.3 Needle Bending and Leakage

Analysis will be performed using a binary logistic regression with random subject effect and fixed pen needle type effect, pair order effect, PN order effect within pair and abdomen site effect. The average difference in percentage of occurrence with BD PN and Terumo PN will be calculated with 95% confidence interval and assessed for statistical significance. The upper bound of the confidence interval will be compared to 0: superiority will be concluded given that the upper bound of the 95% confidence interval for the difference in proportions is < 0%.

DBC-18PENDL01 



```
contrast estimate SE df asymp.LCL asymp.UCL BD Nano - Terumo -0.00000001142909 2759378 NA -5408282 5408282
```

Confidence level used: 0.95

# 6.2.4 Analysis of Exploratory Objectives (Delivery time, Total injection time, Needle Breaking, and Non-Comparative Questionnaire)

#### 6.2.4.1 Delivery time and Total injection time

A mixed effect model will be used (fixed effects of pen needle type, abdomen site, order of pair, order of pen needle within pair and random subject effect) to estimate average difference (BD PN - Terumo PN) in delivery time and total injection time. A Box-Cox transformation might be used to normalize the data if necessary. The upper bound of the confidence interval will be compared to 0: superiority will be concluded given that the upper bound of the 95% interval for the average difference is < 0 seconds.

#### 6.2.4.2 Needle Breaking

The number and proportion of needle breaking occurrence for each pen needle type will be summarized. In addition, a 95% confidence interval for difference in proportions will be calculated using the score method for independent proportions.

## 6.2.4.3 Non-Comparative Questionnaire

All the responses from Non-Comparative Questionnaire will be summarized with number and percentage of each option.

# 7 Safety Analysis

Data listings will be provided for any adverse events and serious adverse events in Appendix. The events will also be summarized descriptively per pen needle type. No safety analysis is planned.

DBC-18PENDL01 



# 8 Example Reports

This section provide examples of tables and graphical representations that will be provided in the study statistical report. These table examples were generated using the sample data available from the data base test framework which do not provide an exhaustive or representative example of the values and levels that will be obtained in the study. They are intended to provide illustrative examples of the tables and figures that will be included in the final statistical analysis report.

# 8.1 Study Execution

The number of subjects enrolled, randomized, withdrawn, who completed and who are excluded will be provided as in Table 1. More details on specific data may be provided in Summary Statistics and Appendix.

## 8.1.1 Analysis Population Set(s)

Table 1: (PP) Population Disposition (Example only)

| Subject.Population | N | Comments |
|----------------------------------------|-----|--------------|
| Subjects Enrolled | 252 | none |
| Subjects who did not meet I/E Criteria | 6 | none |
| Subjects Randomized | 245 | none |
| Subjects Withdrawn | 5 | none |
| Subjects who Completed the Study | 240 | none |
| Subjects Excluded from Analysis | 1 | Give Reasons |

#### 8.1.2 Data Exclusions

All exclusions will be listed with reason(s) for exclusion.

DBC-18PENDL01 



#### 8.1.3 Executive Summary

A high level summary will be provided for each objective/endpoint (example below).

# Primary Objective (examples only):

• Injection Pain: The lower bound of the CI for the average relative pain comparison between BD Nano™ PRO and Terumo Nanopass<sup>®</sup> met both non-inferiority and superiority criteria.

## Secondary Objectives (examples only):

- *Injection force*: The lower bound of the CI for the average difference in rating of BD Nano<sup>™</sup> PRO and Terumo Nanopass<sup>®</sup> injection force met the superiority criterion.
- Needle Bending: The upper bound of the CI for the average difference in percentage of needle bending occurrence with BD Nano<sup>TM</sup> PRO and Terumo Nanopass<sup>®</sup> met the superiority criterion.
- Leakage: The upper bound of the CI for the average difference in percentage of leakage occurrence with BD Nano<sup>TM</sup> PRO and Terumo Nanopass<sup>®</sup> met the superiority criterion.

In addition, a summary table for all primary and secondary objectives will be presented as in Table 2 (Example only). A blue check mark ( $\checkmark$ ) indicates that the acceptance criterion is met, while a red X mark ( $\stackrel{\triangleright}{\times}$ ) indicates that the acceptance criterion is not met.

Table 2: Results Summary of primary and secondary objectives (Example only)

| Objective | |
|----------------------------------|----------|
| Primary Objective | |
| Injection Pain (Non-inferiority) | × |
| Injection Pain (Superiority) | × |
| Secondary Objective | |
| Injection force | <b>✓</b> |
| Needle Bending | <b>✓</b> |
| Leakage | <b>✓</b> |

# 8.2 Analysis and Results

#### 8.2.1 Injection Pain

Summary statistics for the VAS scale will be presented as in Table 3.

The results for average relative VAS Score for BD  $Nano^{TM}$  PRO vs Terumo  $Nanopass^{\textcircled{R}}$  will be evaluated as presented in Table 4.

Table 3: Summary Statistics for observed 150mm Relative VAS Scores (Example only)

| | N | Mean | Std. Dev. | Mean 95% CI | Median | Median 95% CI | Range |
|---|---|---|---|---|---|---|---|
| Injection pain | 13 | 12.12 | 44.00 | (-74.13, 98.36) | 15.00 | (-71.25, 101.25) | -75, 67.5 |

DBC-18PENDL01 



Table 4: Fitted Average Relative VAS score for BD Nano vs Terumo Nanopass (Example only)

| | Fitted Mean | CI | Non-Inferiority | Superiority |
|---|---|---|---|---|
| | | | Conclusion (Lower | Conclusion (Lower |
| | | | bound $CI > -10$ ) | bound $CI > 0$ ) |
| Injection pain | 28.3 | (17.1, 39.4) | TRUE | TRUE |



Figure 2: Distribution of relative VAS scores with average and confidence interval per pen needle group and overall. Positive scores indicate that BD Next was preferred and negative scores indicate that the Current/Assigned PN was preferred. Note: This example graph comes from a study with different PN. Results for this study will reflect BD Nano performance.

DBC-18PENDL01 



# 8.2.2 Injection force

The distribution of the ratings of injection force will be presented as in Table 5 and Figure 3. Summary statistics for the ratings of injection force will be presented as in Table 6.

The results of average ratings will be evaluated as presented in Table 7.

Table 5: Distribution of injection force ratings (Example only)

| ů ( | 1 0 / |
|-----------------------------------------------------|-------------|
| Rating | n (%) |
| -2 (Terumo Nanopass significantly less thumb force) | |
| -1 (Terumo Nanopass slightly less thumb force) | 66 (20.0%) |
| 0 (No Difference) | 66 (20.0%) |
| 1 (BD Nano slightly less thumb force) | 66 (20.0%) |
| 2 (BD Nano significantly less thumb force) | 66 (20.0%) |
| Total | 330 |
| All Rating: >0 | 132 (43.9%) |

Table 6: Summary Statistics for observed ratings of injection force (Example only)

| | N | Mean | Std. Dev. | Mean 95% CI | Median | Median 95% CI | Range |
|---|---|---|---|---|---|---|---|
| Rating of injection force | 330 | 1.4 | 0.1 | [-0.1, 2] | 1.5 | [-0.1, 2] | -2, 2 |

#### Summary for observed ratings of injection force



Figure 3: Observed ratings of injection force (Example only)

DBC-18PENDL01 



Table 7: Fitted average ratings of injection force (Example only)

| | Mean | CI | Superiority Conclusion (Lower bound $CI > 0$ ) |
|---|---|---|---|
| Injection force | 1.30 | [-0.1, 2] | Fail |

The difference in percentage of responses with a preference for BD vs Terumo needle will be presented as in Table 8.

Table 8: Difference in Percentage of responses with a preference for BD Nano vs Terumo Nanopass (Example only)

| percentage of responses with a | percentage of responses with | Difference in Percentage (BD | 95% CI for Difference |
|---|---|---|---|
| preference for BD Nano | a preference for Terumo | Nano - Terumo Nanopass) | |
| | Nanopass | | |
| 45.5% | 40.0% | 4.5% | [2%, 6.8%] |

## 8.2.3 Needle Bending

Summary statistics for needle bending will be presented as in Table 9.

The results of difference in percentage of needle bending will be evaluated as presented in Table 10.

Table 9: Observed percentage of Needle Bending (Example only)

| Pen Needle | Needle bending | 95% CI |
|-----------------|-------------------|-------------|
| BD Nano | 4/330 (1.2%) | [0.1%, 2%] |
| Terumo Nanopass | $4/330 \ (1.2\%)$ | [0.1%, 2%] |

Table 10: Difference in Percentage of Needle Bending (Example only)

| Comparison | Difference in Percentage of Needle bending based on modeling analysis. | 95% CI for Difference |
|---|---|---|
| BD Nano vs Terumo Nanopass | -1.2% | [-2%, 0.8%] |

#### 8.2.4 Leakage from Injection Site

Summary statistics for leakage from injection site will be presented as in Table 11. The distribution of leakage from injection site will be presented as in Figure 4.

The leakage on a binary scale will also be presented and analyzed as in Section 8.2.3.

Table 11: Summary Statistics for leakage from injection site (Example only)

| Pen needle | N | Mean | Std. Dev. | Median | Range |
|------------|---|------|-----------|--------|----------------|
| BD Nano | 3 | 0.02 | 0.02 | 0.02 | 0.0112, 0.0298 |

 $[1]\ 0.0276[1]\ 0.01903506$ 

DBC-18PENDL01 





Figure 4: Leakage from the Injections per Pen Needle Type. The blue like represents the threshold for leakage (0.015g).

DBC-18PENDL01 



# 8.2.5 Exploratory Objectives

Patient end needle breaking will be summarized as in Section 8.2.3.

Summary statistics for delivery time and total injection time will be presented as in Table 12. The average difference (BD PN - Terumo PN) in delivery time and total injection time will be evaluated as presented in Table 13.

Table 12: Summary Statistics for delivery time (Example only)

| Pen Needle | N | SD | Mean | Median | Range |
|-----------------|----|-------|--------|--------|------------|
| BD Nano | 31 | 40.52 | 142.03 | 142.00 | 90,274 |
| Terumo Nanopass | 31 | 63.90 | 165.84 | 140.00 | $91,\!362$ |

Table 13: Mean difference of Delivery time and Total injection time with confidence interval (reciprocal of number of seconds). The last column indicates whether superiority was met or not. (Example only)

| | Mean difference | 95% Lower bound | P value | Lower bound >0 (Superiority) |
|---|---|---|---|---|
| Delivery time | 0.000739 | -0.000180 | 0.113 | Fail |
| Total injection time | 0.000452 | -0.000180 | 0.279 | Fail |

# 8.3 Demographics and Diabetes History

Table 14: Subject Demographics (Example only)

| | J 0 1 | \ 1 |
|------|-------------------|------------|
| Char | acteristic | Results |
| Geno | ler | |
| | Female | 94 (50.8%) |
| | Male | 91~(49.2%) |
| Age | | |
| | Mean | 55.8 |
| | 95% Mean CI | 53.9, 57.7 |
| | SD | 13.0 |
| | Min, Max | 20, 76 |
| | Observation Count | 183 |
| | Missing Count | 2 |
| | Total Count | 185 |

Table 15: Distribution of Type of Diabetes (Example only)

| Characteristic | Results |
|----------------|-------------|
| Diabetes Type | |
| Type II | 152~(84.4%) |
| Type I | 28~(15.6%) |
| Missing | 2 |

DBC-18PENDL01 



Table 16: Diabetes History (Example only)

| Characteristic | Results |
|-------------------------------|-----------------|
| Diagnosed year | |
| Mean | 14.2 |
| 95% Mean CI | 12.8, 15.6 |
| $\operatorname{SD}$ | 9.4 |
| Min, Max | 1, 54 |
| Total Count | 182 |
| Injection Times per day | |
| once | 74 (40.7%) |
| four | 36 (19.8%) |
| twice | $31\ (17.0\%)$ |
| five or more | 19~(10.4%) |
| NA - injects non-insulin only | 11~(~6.0%) |
| three | 11~(~6.0%) |
| Pen needle used | |
| BD Nano 32Gx4mm | 66~(36.5%) |
| NovoFine 32Gx6mm | 33~(18.2%) |
| Other 32G | $24\ (13.3\%)$ |
| Other 31Gx5mm | $22\ (12.2\%)$ |
| NovoTwist 32Gx5mm | $20 \ (11.0\%)$ |
| NovoFine Plus 32Gx4mm | 14~(~7.7%) |
| Owen Mumford PenTips 32Gx4mm | 2 (1.1%) |
| Missing | 1 |
| Injection site used | |
| Abdomen | 158~(87.3%) |
| Thigh | 14~(~7.7%) |
| $\operatorname{Arm}$ | 7 ( 3.9%) |
| Buttocks | 1~(~0.6%) |
| Other | 1~(~0.6%) |
| Missing | 1 |

DBC-18PENDL01 



# 9 Appendix

## 9.1 Discontinued Data

The Table 17 shows the detailed list of discontinued subjects.

Table 17: Details of Discontinued Subjects (Example only)

| Subject ID | Completion Date | Discontinuation Time | Reason for Discontinuation | Details |
|---|---|---|---|---|
| R003 | January 3, 2018 | After initiation of study | Other | Subject decided not con- |
| | | procedure/ intervention | | tinue to participate |
| R067 | February 7, 2018 | Before any study proce- | Did not meet criteria | |
| | | dure/ intervention | (Screen Failure) | |
| R114 | February 19, 2018 | After initiation of study | Administrative Issue | Detail of reason for discon- |
| | | procedure/ intervention | | tinuation |

# 9.2 Missing Data

All the Missing data will be listed.

## 9.3 Adverse Events

Data listings will be provided for any adverse events and serious adverse event in Table 18. Adverse events will be summarized descriptively by pen needle in Table 19 and 20.

Table 18: Data listing for adverse events (Example only)

| Random | PN Used | Seriousness | Severity | Relation to | Contribution | Relation to | Description |
|---|---|---|---|---|---|---|---|
| ID | | | | product | of product | protocol | |
| | | | | | malfunction | | |
| R055 | BD Nano | Serious | Moderate | Related | Yes | Not related | adverse event to be described |
| R001 | Terumo | Serious | Mild | Unlikely re- | No | Possibly re- | adverse event to be described |
| | Nanapass | | | lated | | lated | |
| R099 | Terumo | Serious | Severe | Possibly re- | Yes | related | adverse event to be described |
| | Nanapass | | | lated | | | |

Table 19: Summary of Adverse Events: Relationship to product (Example only)

| | | | | | ` - | |
|---|---|---|---|---|---|---|
| Pen Needle | Number of | Number of | Not related | Unlikely re- | Possibly re- | Related |
| | events | Subjects | | lated | lated | |
| BD Nano | 5 | 2 | 2 | 1 | 1 | 1 |
| BD Nano | 0 | 0 | 0 | 0 | 0 | 0 |
| BD Nano | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 3 | 2 | 1 | 0 | 2 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |

DBC-18PENDL01 



Table 20: Summary of Adverse Events: Relationship to protocol / procedure (Example only)

| Pen Needle | Number of | Number of | Not related | Unlikely re- | Possibly re- | Related |
|---|---|---|---|---|---|---|
| | events | Subjects | | lated | lated | |
| BD Nano | 5 | 2 | 2 | 1 | 1 | 1 |
| BD Nano | 0 | 0 | 0 | 0 | 0 | 0 |
| BD Nano | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 3 | 3 | 0 | 1 | 0 | 2 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 3 | 2 | 1 | 0 | 2 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |
| Terumo Nanapass | 0 | 0 | 0 | 0 | 0 | 0 |

DBC-18PENDL01 